CLINICAL TRIAL: NCT01964040
Title: Perineural Dexmedetomidine as an Adjuvant to Bupivacaine-induced Ultrasound-guided Femoral Nerve Block.
Brief Title: Perineural Dexmedetomidine and Femoral Nerve Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Collaborators: anesthesia department (Ambiguous); faculty of medicine (Ambiguous)
Responsible Party: Principal Investigator, Abeer Ahmed, lecturer of anesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: N-38-2013
Record Dates: First submitted 2013-09-26; First posted 2013-10-17 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-10

CONDITIONS: Onset and Duration of Sensory and Motor Block of Femoral Nerve,; Visual Analogue Pain Scores,; Time to First Request of Rescue Analgesics,; Total Morphine Consumption in 24 Hours
Keywords: femoral nerve block; peri-neural dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- group B: control bupivacaine group (Placebo Comparator): Patient in this group will receive 25 ml bupivacaine 0.5% plus 0.5 ml normal saline peri-neurally and 0.5 ml subcutaneous normal saline.
  Interventions: Drug: peri-neural dexmedetomidine as adjuvant to bupivacaine in femoral nerve block
- Group B-peri-DEX: Peri-neural Dexmedetomidine (Experimental): Patients in this group will receive 25 ml of 0.5% bupivacaine plus 0.5 ml (50 microgram) Dexmedetomidine peri-neurally and 0.5 ml subcutaneous normal saline
  Interventions: Drug: peri-neural dexmedetomidine as adjuvant to bupivacaine in femoral nerve block
- Group B-sys-DEX:Systemic Dexmedetomidine (Active Comparator): Patients in this group will receive 25 ml bupivacaine plus 0.5 ml saline peri-neurally and 0.5 ml (50 microgram) subcutaneous Dexmedetomidine.
  Interventions: Drug: peri-neural dexmedetomidine as adjuvant to bupivacaine in femoral nerve block

INTERVENTIONS:
Drug: peri-neural dexmedetomidine as adjuvant to bupivacaine in femoral nerve block — ultrasound quided femoral nerve block with injection of 15 ml bupivacaine 0.5% perineurally with 0.5 ml dexmedetomidine (50 microgram) either perineurally or subcutaneously.
  After adequate assessment of femoral nerve block, patients will be transferred to the operating room to receive a standard general anesthesia

SUMMARY:
The duration of sensory block after single dose of long acting local anesthetics is not sufficient to avoid the postoperative use of opioids. Alpha-2 adrenoceptor agonists such as clonidine have been shown to increase the duration of peripheral nerve block. Dexmedetomidine is a more potent and selective α-2-adrenoceptor compared to clonidine. To the best of our knowledge, the use of Dexmedetomidine as adjuvant to local anesthetic was not previously reported for femoral nerve block.

ELIGIBILITY:
Inclusion Criteria:

* all patients with ASA physical status I or II, scheduled for diagnostic knee arthroscopy

Exclusion Criteria:

* Patients who are refusing regional block, patients with diabetic peripheral neuropathy, renal or hepatic dysfunction, inflammation or infection at the puncture site, and history of allergic reaction to study medications

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2013-08; Primary Completion 2013-12 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure of this study will be the change of sensory block over time. | intraoperatively every 5 minutes for the first 30 minutes of the operation, then postoperatively every 2 hours for 24hours
  Over a period of 30 min after injection of the study medications, a blinded investigator will assess sensory block with pinprick test using a 3-point scale: 0 ═ complete loss of sensation, 1 ═ partial loss of sensation and 2 ═ normal sensation (10). Pinprick test will be done in comparison to the contralateral area at the sensory distribution of the femoral nerve

SECONDARY OUTCOMES:
onset of motor and sensory block | up to 30 minutes after the end of injection
  The onset time of sensory and motor block will be: "the time elapsed between the end of injection and the development of complete block (score of 0 at all dermatomes or no movement of the quadriceps muscle.

OTHER OUTCOMES:
duration of motor block | interval between time of injection and complete motor power recover
  The duration of motor block will be defined as: "the time interval between the end of injection and the complete recovery of motor power of the quadriceps muscle)".
Visual analogue pain scores (resting and dynamic) and Richmond Agitation-Sedation Score (RASS) ( | 2hours post operative and for 24hours
  Visual analogue pain scores (resting and dynamic) and Richmond Agitation-Sedation Score (RASS) (12) will be assessed at 2, 4, 6, 8, 12, 16, and 24 hours postoperatively
time of 1st request of rescue analgesia | over the poatoperative 24hours
  The time to the first request of rescue postoperative analgesic will be: "the time interval between the onset of successful sensory block and the first request to postoperative analgesia"

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesia department-faculty of medicine-Cairo University, Cairo, Cairo Governorate, Egypt